CLINICAL TRIAL: NCT00595894
Title: RA Comorbidity: Bone Health in Men and African Americans
Brief Title: Rheumatoid Arthritis Comorbidity: Bone Health in Men and African Americans
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0028-03-ET; 5K23AR050004-04 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; African Americans; osteopenia; osteoporosis; bone mineral density
MeSH Terms: conditions — Arthritis, Rheumatoid; Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Baseline sera and DNA collected
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 CLEAR participants - African Americans with early rheumatoid arthritis: CLEAR enrollees include African American patients with early rheumatoid arthritis, as defined using ACR criteria
- 2 VARA participants - male veterans with established rheumatoid arthritis: VARA enrollees will include male veterans with established RA diagnosed using ACR criteria

SUMMARY:
The objective of the proposed study is to assess bone health and determinants of bone health among select subpopulations of rheumatoid arthritis patients.

DETAILED DESCRIPTION:
The overall hypothesis of this study is that osteopenia and/or osteoporosis are common among African Americans and men with rheumatoid arthritis and there are identifiable genetic and environmental factors contributing to the pathogenesis of bone loss in these groups.

The Specific Aims of the study are to:

1. Determine baseline hip and lumbar spine bone density (BMD) values and osteopenia/osteoporosis prevalence among African American men and women with early RA and among male veterans with established RA.
2. Identify environmental factors and candidate alleles, which confer increased risk of reduced baseline BMD loss over time among African American men and women with early RA and among male veterans with established RA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rheumatoid arthritis per ACR guidelines

Exclusion Criteria:

* Patients with diagnosis > 2yrs (CLEAR study)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLEAR enroll African American RA patients from 4 core academic centers in the Southeast U.S. VARA enroll RA patientss from participating VA medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 1745 (Actual)
Dates: Start 2004-07-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | baseline and at 5 years disease
  Bone mineral density (BMD) test measures calcium and other minerals in bone. Bones containing more minerals are denser, so they tend to be stronger and less likely to break.

CONTACTS AND LOCATIONS:
Overall Officials: Ted R Mikuls, MD, MSPH, Principal Investigator — University of Nebraska
Locations (1):
- Omaha Veteran's Affairs Medical Center, Omaha, Nebraska, United States

REFERENCES:
- See also: National Institute of Health — http://www.nih.gov